CLINICAL TRIAL: NCT01050374
Title: Gaps in Helminth Control: Safety and Efficacy of Drug Combinations. Praziquantel Study
Brief Title: Safety and Efficacy of Drug Combinations Against Schistosomiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Responsible Party: Harriet Namwanje Principal Investigator, Vector control division, Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AO.UGA.PZQ; DBL-CHRD
Record Dates: First submitted 2008-01-23; First posted 2010-01-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Parasitic Diseases
MeSH Terms: conditions — Parasitic Diseases | interventions — Albendazole; Praziquantel; Mebendazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): albendazole + praziquantel
  Interventions: Drug: albendazole + praziquantel
- 2 (Active Comparator): mebendazole + praziquantel
  Interventions: Drug: mebendazole + praziquantel

INTERVENTIONS:
Drug: albendazole + praziquantel — albendazole (400 mg one dose) + praziquantel (40 mg/kg body weight)
  Arms: 1
Drug: mebendazole + praziquantel — mebendazole (500 mg one dose) + praziquantel (40 mg/kg body weight)
  Arms: 2

SUMMARY:
This randomised, controlled, double-blinded clinical study investigates the safety and efficacy of MBD in combination with PZQ in the treatment of SCH and STH in children aged 1-15 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Those with an age of 1-15 years of age
* Are infected with schistosomiasis and soil-transmitted helminthiasis
* Whose parent consent and who are willing to participate

Exclusion Criteria:

* Those with acute and chronic diseases other than schistosomiasis and soil-transmitted helminthiasis
* Those with a history of any serious adverse drug reactions

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 650 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment | 6 weeks

SECONDARY OUTCOMES:
Record of adverse reactions | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Vector Control Division, Kampala, Uganda